CLINICAL TRIAL: NCT02397096
Title: A Phase III Multicenter, Open-Label, Randomized Study to Evaluate a Switch to MK-1439A in HIV-1-Infected Subjects Virologically Suppressed on a Regimen of a Ritonavir-boosted Protease Inhibitor and Two Nucleoside Reverse Transcriptase Inhibitors (NRTIs)
Brief Title: Safety and Efficacy of a Switch to Doravirine, Tenofovir, Lamivudine (MK-1439A) in Human Immunodeficiency Virus (HIV-1)-Infected Participants Virologically Suppressed on an Anti-retroviral Regimen in Combination With Two Nucleoside Reverse Transcriptase Inhibitors (MK-1439A-024)
Acronym: DRIVE-SHIFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1439A-024; MK-1439A-024 (Other: MSD ID); 2014-005550-18 (EudraCT Number)
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — doravirine; Tenofovir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate Switch to Doravirine, Tenofovir, Lamivudine (Experimental): Participants receiving continuous antiretroviral therapy with a ritonavir- or cobicistat-boosted protease inhibitor (atazanavir, darunavir, or lopinavir) or cobicistat-boosted elvitegravir or a non nucleoside reverse transcriptase inhibitor (NNRTI) (specifically, efavirenz, nevirapine, or rilpivirine) in combination with 2 NRTIs for >=6 months with undetectable HIV-1 RNA will switch on Day 1 to doravirine, tenofovir, lamivudine single tablet by mouth once daily for 48 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions
  Interventions: Drug: Doravirine, Tenofovir, Lamivudine; Drug: Baseline regimen of ritonavir- or cobicistat-boosted protease inhibitor; Drug: Baseline regimen of cobicistat-boosted elvitegravir; Drug: Baseline regimen of a non-nucleoside reverse transcriptase inhibitor; Drug: Baseline regimen of two nucleoside reverse transcriptase inhibitors
- Delayed Switch to Doravirine, Tenofovir, Lamivudine (Active Comparator): Participants receiving continuous antiretroviral therapy with a ritonavir- or cobicistat-boosted protease inhibitor (atazanavir, darunavir, or lopinavir) or cobicistat-boosted elvitegravir or a NNRTI (specifically, efavirenz, nevirapine, or rilpivirine) in combination with 2 NRTIs for >=6 months with undetectable HIV-1 RNA will continue on this therapy until Week 24, at which time they will switch to doravirine, tenofovir, lamivudine single tablet by mouth once daily for 24 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions
  Interventions: Drug: Doravirine, Tenofovir, Lamivudine; Drug: Baseline regimen of ritonavir- or cobicistat-boosted protease inhibitor; Drug: Baseline regimen of cobicistat-boosted elvitegravir; Drug: Baseline regimen of a non-nucleoside reverse transcriptase inhibitor; Drug: Baseline regimen of two nucleoside reverse transcriptase inhibitors

INTERVENTIONS:
Drug: Doravirine, Tenofovir, Lamivudine — Single tablet containing MK-1439 (doravirine) 100 mg, lamivudine 300 mg, and tenofovir disoproxil fumarate 300 mg
  Other Names: Doravirine (PIFELTRO™); Doravirine/Lamivudine/Tenofovir disoproxil fumarate (DELSTRIGO™); MK-1439A
Drug: Baseline regimen of ritonavir- or cobicistat-boosted protease inhibitor — Baseline regimen of antiretroviral therapy with a ritonavir- or cobicistat-boosted protease inhibitor (atazanavir, darunavir, or lopinavir) administered according to the product circular
Drug: Baseline regimen of cobicistat-boosted elvitegravir — Baseline regimen of antiretroviral therapy with cobicistat-boosted elvitegravir administered according to the product circular
Drug: Baseline regimen of a non-nucleoside reverse transcriptase inhibitor — Baseline regimen of antiretroviral therapy with a NNRTI (efavirenz, nevirapine, or rilpivirine) administered according to the product circular
Drug: Baseline regimen of two nucleoside reverse transcriptase inhibitors — Baseline regimen of antiretroviral therapy with two NRTIs administered according to the product circular

SUMMARY:
The multicenter, open label, randomized study will evaluate the safety and efficacy of a switch to MK-1439A (MK-1439 [doravirine] plus lamivudine and tenofovir disoproxil fumarate) in HIV-1-infected participants virologically suppressed on a protocol-specified antiretroviral regimen. The primary hypothesis is that a switch to doravirine, tenofovir, lamivudine will be non-inferior to continuation of the regimen at Screening for 24 weeks, as assessed by the proportion of participants maintaining HIV-1 ribonucleic acid (RNA) <50 copies/mL. The Base Study results will be based on the first 48 weeks of this ongoing study.

DETAILED DESCRIPTION:
Three optional study extensions are planned. Study Extension 1 will evaluate safety of the switch to doravirine, tenofovir, lamivudine for an additional 2 years beyond the Base Study. Study Extensions 2 and 3 will evaluate safety of the switch to doravirine, tenofovir, lamivudine until doravirine, tenofovir, lamivudine becomes locally available, or 4 years beyond Study Extension 1, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria include, but are not limited to:

* Have plasma Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) levels below the limit of quantification (BLoQ) (<40 copies/mL by the Abbott RealTime HIV-1 Assay as determined by the central laboratory) at the screening visit.
* Receiving antiretroviral therapy with a ritonavir- or cobicistat-boosted protease inhibitor (atazanavir, darunavir, or lopinavir) or cobicistat-boosted elvitegravir or a NNRTI (specifically, efavirenz, nevirapine, or rilpivirine) in combination with 2 Nucleoside Reverse Transcriptase Inhibitor (NRTIs) (and no other antiretroviral therapy) continuously for >= 6 months.
* Receiving first or second retroviral regimen (participants receiving a NNRTI at Screening must be on their first retroviral regimen)
* No history of using an experimental NNRTI
* Has a genotype prior to starting his/her initial antiretroviral regimen and no known resistance to any of the study agents
* Not receiving lipid lowering therapy or on a stable dose of lipid lowering therapy at the time of enrollment
* Has the following laboratory values at screening within 30 days prior to the treatment phase of this study: Alkaline phosphatase ≤ 3.0 x upper limit of normal (ULN), Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤ 5.0 x ULN, and Hemoglobin ≥9.0 g/dL (if female) or ≥10.0 g/dL (if male)
* Has a calculated creatinine clearance at the time of screening ≥ 50 mL/min, based on the Cockcroft-Gault equation
* Male or female participant not of reproductive potential or, if of reproductive potential, agrees to avoid becoming pregnant or impregnating a partner while receiving study drug and for 14 days after the last dose of study drug by complying with one of the following: 1) practice abstinence from heterosexual activity, or 2) use acceptable contraception during heterosexual activity
* For inclusion in Study Extension 1 (optional): completed the Week 48 visit; considered to have derived benefit from study participation up to Week 48; considered to be a clinically appropriate candidate for an additional 2 years treatment with study drug
* For inclusion in Study Extension 2 (optional): completed the Week 144 visit; considered to have derived benefit from study participation up to Week 144; considered to be a clinically appropriate candidate for an additional 2 years treatment with study drug
* For inclusion in Study Extension 3 (optional): completed the Week 240 visit; considered to have derived benefit from study participation up to Week 240; considered to be a clinically appropriate candidate for an additional 2 years treatment with study drug

Exclusion Criteria:

Exclusion Criteria include, but are not limited to:

* Uses recreational or illicit drugs or has a recent history of drug or alcohol abuse or dependence
* Received treatment for a viral infection other than HIV-1, such as hepatitis B, with an agent that is active against HIV-1 such as adefovir, emtricitabine, lamivudine, or tenofovir
* Has documented or known resistance to study drugs including doravirine, lamivudine, and/or tenofovir
* Participated in a study with an investigational compound or device within 30 days or anticipates doing so during the course of this study
* Used systemic immunosuppressive therapy or immune modulators within 30 days or anticipates needing them during the course of this study (short courses of corticosteroids will be allowed)
* Current, active diagnosis of acute hepatitis due to any cause (participants with chronic hepatitis B and C may enter the study as long as they fulfill all entry criteria, have stable liver function tests, and have no significant impairment of hepatic function)
* Has evidence of decompensated liver disease or has liver cirrhosis and a Child-Pugh Class C score or Pugh-Turcotte score >9
* Pregnant, breastfeeding, or expecting to conceive at any time during the study
* Female and is expecting to donate eggs or male and is expecting to donate sperm during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Orkin C, Koethe JR, Kumar PN, Sklar P, Xu ZJ, Plank RM, Greaves W, Lahoulou R. Factors Associated With Weight Change After Continuing or Switching to a Doravirine-based Regimen. Open Forum Infect Dis. 2025 Nov 20;12(11):ofaf639. doi: 10.1093/ofid/ofaf639. eCollection 2025 Nov. PMID 41280318
- [Derived] Walmsley SL, Kumar PN, Orkin C, Thompson M, Squires K, Xu ZJ, Greaves W, Plank RM, Whiteside Y, Lahoulou R. Efficacy and Safety of Doravirine-based Regimens by Sex and Race: Long-term Results From Three Phase 3 Clinical Trials. Open Forum Infect Dis. 2025 Jul 16;12(7):ofaf356. doi: 10.1093/ofid/ofaf356. eCollection 2025 Jul. PMID 40672760
- [Derived] Kumar P, Johnson M, Molina JM, Rizzardini G, Cahn P, Bickel M, Wan H, Xu ZJ, Morais C, Sklar P, Greaves W; DRIVE-SHIFT Study Group. Brief Report: Switching to DOR/3TC/TDF Maintains HIV-1 Virologic Suppression Through Week 144 in the DRIVE-SHIFT Trial. J Acquir Immune Defic Syndr. 2021 Jun 1;87(2):801-805. doi: 10.1097/QAI.0000000000002642. PMID 33633036
- [Derived] Vaddady P, Kandala B, Yee KL. Population Pharmacokinetic and Pharmacodynamic Analysis To Evaluate a Switch to Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate in People Living with HIV-1. Antimicrob Agents Chemother. 2020 Oct 20;64(11):e00590-20. doi: 10.1128/AAC.00590-20. Print 2020 Oct 20. PMID 32868326
- [Derived] Johnson M, Kumar P, Molina JM, Rizzardini G, Cahn P, Bickel M, Mallolas J, Zhou Y, Morais C, Kumar S, Sklar P, Hanna GJ, Hwang C, Greaves W; DRIVE-SHIFT Study Group. Switching to Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (DOR/3TC/TDF) Maintains HIV-1 Virologic Suppression Through 48 Weeks: Results of the DRIVE-SHIFT Trial. J Acquir Immune Defic Syndr. 2019 Aug 1;81(4):463-472. doi: 10.1097/QAI.0000000000002056. PMID 30985556
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26154&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 852 participants screened, 673 were randomized to study treatment, and 670 were treated. There were 122 global study sites utilized.
Groups:
- Immediate Switch Group (ISG): Participants received continuous antiretroviral therapy with a ritonavir- or cobicistat-boosted protease inhibitor (atazanavir, darunavir, or lopinavir) or cobicistat-boosted elvitegravir or a non nucleoside reverse transcriptase inhibitor (NNRTI) (specifically, efavirenz, nevirapine, or rilpivirine) in combination with 2 (nuceloside/nucleotide reverse transcriptase inhibitors) NRTIs for >=6 months with undetectable HIV-1 RNA switched on Day 1 to MK-1439A single tablet by mouth once daily for 48 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions.
- Delayed Switch Group (DSG): Participants received continuous antiretroviral therapy with a ritonavir- or cobicistat-boosted protease inhibitor (atazanavir, darunavir, or lopinavir) or cobicistat-boosted elvitegravir or a NNRTI (specifically, efavirenz, nevirapine, or rilpivirine) in combination with 2 NRTIs for >=6 months with undetectable HIV-1 RNA continued on this therapy until Week 24, at which time they switched to MK-1439A single tablet by mouth once daily for 24 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions.
Period: Day 1 to Week 24
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Started | 450 | 223
Treated | 447 | 223
Completed | 427 | 209
Not Completed | 23 | 14
Not completed — Adverse Event | 7 | 1
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 3 | 4
Not completed — Physician Decision | 2 | 3
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Randomized, not treated | 3 | 0
Period: Week 24 to Week 48
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Started | 427 | 209
Completed | 407 | 202
Not Completed | 20 | 7
Not completed — Adverse Event | 6 | 2
Not completed — Lack of Efficacy | 5 | 1
Not completed — Non-Compliance With Study Drug | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 2 | 0
Period: Study Extension 1
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Started | 398 (Number started refers only to participants completing Base Study volunteering to continue to Study Extension Part 1.) | 202
Completed | 357 | 179
Not Completed | 41 | 23
Not completed — Adverse Event | 7 | 5
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 2 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Non-compliance with study drug | 3 | 0
Not completed — Physician Decision | 4 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 21 | 7
Period: Study Extension 2
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Started | 303 (Number started refers only to participants completing Base Study and Study Extension Part 1 and volunteering to continue to Study Extension Part 2.) | 154 (Number started refers only to participants completing Base Study and Study Extension Part 1 and volunteering to continue to Study Extension Part 2.)
Completed | 129 | 78
Not Completed | 174 | 76
Not completed — Adverse Event | 3 | 3
Not completed — Availability of study medication locally | 152 | 64
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Physician Decision | 2 | 5
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 10 | 3
Period: Study Extension 3
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Started | 84 (Number started refers only to participants completing Base Study, Study Extension Part 1, Study Extension Part 2 and volunteering to continue to Study Extension Part 3.) | 43 (Number started refers only to participants completing Base Study, Study Extension Part 1, Study Extension Part 2 and volunteering to continue to Study Extension Part 3.)
Completed | 69 | 39
Not Completed | 15 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Availability of study medication locally | 11 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG) | Total
Number analyzed (Participants) | 450 | 223 | 673
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (10.1) | 43.7 (10.6) | 43.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 29 | 104
  Male | 375 | 194 | 569
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 98 | 43 | 141
  Not Hispanic or Latino | 347 | 177 | 524
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 17 | 8 | 25
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 56 | 34 | 90
  White | 346 | 168 | 514
  More than one race | 25 | 11 | 36
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) <50 Copies/mL
Description: The percentage of participants in each arm achieving HIV-1 RNA levels <50 copies/mL was determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach and all missing data were considered treatment failures, regardless of the reason.
Time Frame: Immediate Switch to MK-1439A arm: Week 48; Delayed Switch to MK-1439A arm: Week 24
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 447 | 223
Percentage of Participants | 90.8 | 94.6
Statistical Analysis 1: Comparison: Immediate Switch Group (ISG) vs Delayed Switch Group (DSG); Test type: Non-Inferiority — Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (DOR/3TC/TDF) once daily (QD) ISG is concluded to be non-inferior to baseline regimen DSG if the lower bound of the 95% CI for the difference in percent response is above -8 percentage points; Treatment Difference = -3.784, 95% CI 2-sided [-7.877 to 0.310] — Stratum-adjusted Mantel-Haenszel method with the difference weighted by the harmonic mean of sample size per arm for each stratum; Superiority of an immediate switch to DOR/3TC/TDF over continuation of the baseline regimen was defined by a lower bound of the two-sided 95% CI for the difference in response rates being greater than zero (contingent upon satisfying the multiplicity criteria)

2. Secondary Outcome: Mean Change From Baseline in Fasting Low-density Lipoprotein Cholesterol (LDL-C)
Description: To evaluate the effect on fasting LDL-C of an immediate switch to DOR/3TC/TDF on Study Day 1 compared with continuation of a ritonavir-boosted, PI-based regimen, as measured by mean change from baseline in each treatment group. The Last Observation Carry Forward (LOCF) approach was applied to missing data and data collected after a participant initiated lipid-modifying therapy.
Time Frame: Baseline and Week 24
Population: All randomized participants in the ritonavir-boosted PI-based regimen who received at least 1 dose of study drug and had a measurement at baseline and had at least one post baseline time point assessed.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Immediate Switch (Ritonavir--boosted, PI-based) Group (ISG): Participants received continuous antiretroviral therapy with a ritonavir-boosted, PI-based regimen for >=6 months with undetectable HIV-1 RNA switched on Day 1 to MK-1439A single tablet by mouth once daily for 48 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions.
- Delayed Switch (Ritonavir-boosted, PI-based) Group (DSG): Participants received continuous antiretroviral therapy with a ritonavir-boosted, PI-based regimen for >=6 months with undetectable HIV-1 RNA continued on this therapy until Week 24, at which time they switched to MK-1439A single tablet by mouth once daily for 24 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions.
Arm/Group | Immediate Switch (Ritonavir--boosted, PI-based) Group (ISG) | Delayed Switch (Ritonavir-boosted, PI-based) Group (DSG)
Number analyzed (Participants) | 256 | 125
mg/dL
  Baseline | 108.82 (34.21) | 109.00 (33.58)
  Change from Baseline | -16.54 (23.10) | -1.94 (25.74)
Statistical Analysis 1: Comparison: Immediate Switch (Ritonavir--boosted, PI-based) Group (ISG) vs Delayed Switch (Ritonavir-boosted, PI-based) Group (DSG); Test type: Other; p < 0.0001, ANCOVA; Treatment Difference = -14.65, 95% CI 2-sided [-18.92 to -10.38] — 95% CIs and 2-sided p-values were calculated from an ANCOVA model with terms for baseline lipid level, use of lipid-lowering therapy at Study Day 1 and treatment

3. Secondary Outcome: Mean Change From Baseline in Fasting Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Serum non-HDL-C was determined after an overnight fast. Change from Baseline was analyzed using ANCOVA models with terms for Baseline lipid level and treatment group. The Last Observation Carry Forward (LOCF) approach was applied for missing data or data collected after modifying lipid lowering therapy.
Time Frame: Baseline and Week 24
Population: All randomized participants who received the ritonavir-boosted PI-based regimen at least 1 dose of study drug and had a measurement at baseline and had at least one post baseline time point assessed.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Immediate Switch (Ritonavir--boosted, PI-based) Group (ISG): Participants receiving continuous antiretroviral therapy with a ritonavir-boosted, PI-based regimen for >=6 months with undetectable HIV-1 RNA switched on Day 1 to MK-1439A single tablet by mouth once daily for 48 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions.
- Delayed Switch (Ritonavir-boosted, PI-based) Group (DSG): Participants receiving continuous antiretroviral therapy with a ritonavir-boosted, PI-based regimen for >=6 months with undetectable HIV-1 RNA continued on this therapy until Week 24, at which time they switched to MK-1439A single tablet by mouth once daily for 24 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions.
Arm/Group | Immediate Switch (Ritonavir--boosted, PI-based) Group (ISG) | Delayed Switch (Ritonavir-boosted, PI-based) Group (DSG)
Number analyzed (Participants) | 266 | 133
mg/dL
  Baseline | 139.14 (42.12) | 137.99 (38.46)
  Change from Baseline | -24.74 (29.26) | -1.31 (28.45)
Statistical Analysis 1: Comparison: Immediate Switch (Ritonavir--boosted, PI-based) Group (ISG) vs Delayed Switch (Ritonavir-boosted, PI-based) Group (DSG); Test type: Other; p < 0.0001, ANCOVA; Treatment Difference = -23.03, 95% CI 2-sided [-28.00 to -18.05] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants Maintaining HIV-1 RNA <50 Copies/mL
Description: as for outcome 1
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 447 | 223
Percentage of Participants | 93.7 | 94.6
Statistical Analysis 1: Comparison: Immediate Switch Group (ISG) vs Delayed Switch Group (DSG); Test type: Non-Inferiority — DOR/3TC/TDF QD ISG is concluded to be non-inferior to baseline regimen DSG if the lower bound of the 95% CI for the difference in percent response is above -8 percentage points; Treatment Difference = -0.877, 95% CI 2-sided [-4.706 to 2.952] — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation (CD4) Cell Counts
Description: The mean change from baseline in CD4 cell counts was assessed using the Observed Failure (OF) approach. With the OF approach, baseline values were carried forward for participants who discontinued due to lack of efficacy. Cell counts were measured and expressed as cells/mm^3, and percent change was then calculated. CD4 cell counts were quantified by a central laboratory using a commercially available assay.
Time Frame: Immediate Switch to MK-1439A arm: Baseline and Week 48; Delayed Switch to MK-1439A arm: Baseline and Week 24
Population: All randomized participants who received at least 1 dose of study drug and had a measurement at baseline and had at least one post baseline time point assessed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 402 | 209
cells/mm^3
  Baseline | 660.5 (293.4) | 655.6 (279.3)
  Change from Baseline | 13.9 (168.1) | 18.0 (157.7)
Statistical Analysis 1: Comparison: Immediate Switch Group (ISG) vs Delayed Switch Group (DSG); Test type: Other; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-31.6 to 23.5] — 95% CIs were calculated based on t-distribution

6. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation (CD4) Cell Counts
Description: The mean change from baseline in CD4 cell counts at Week 48 was assessed using the Observed Failure (OF) approach. With the OF approach, baseline values were carried forward for participants who discontinued due to lack of efficacy. Cell counts were measured and expressed as cells/mm^3, and percent change was then calculated. CD4 cell counts were quantified by a central laboratory using a commercially available assay.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 412 | 209
cells/mm^3
  Baseline | 664.5 (300.7) | 655.6 (279.3)
  Change from Baseline | 5.1 (174.9) | 18.0 (157.7)
Statistical Analysis 1: Comparison: Immediate Switch Group (ISG) vs Delayed Switch Group (DSG); Test type: Superiority; Mean Difference (Final Values) = -12.8, 95% CI 2-sided [-41.1 to 15.4] — 95% Confidence Intervals were based on t-distribution

7. Secondary Outcome: Percentage of Participants Maintaining HIV-1 RNA <40 Copies/mL
Description: The percentage of participants in each arm achieving HIV-1 RNA levels <40 copies/mL was determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach and all missing data were considered treatment failures, regardless of the reason.
Time Frame: Immediate Switch to MK-1439A arm: Week 48; Delayed Switch to MK-1439A arm: Week 24
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 447 | 223
Percentage of Participants | 89.7 | 93.3
Statistical Analysis 1: Comparison: Immediate Switch Group (ISG) vs Delayed Switch Group (DSG); Test type: Other; Treatment Difference = -3.556, 95% CI 2-sided [-7.977 to 0.864] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of Participants Maintaining HIV-1 RNA <40 Copies/mL
Description: To evaluate the immunological effect of an immediate switch to MK -1439A on Study Day 1 compared with continuation of a ritonavir boosted, PI-based regimen, as measured by the proportion of subjects maintaining HIV-1 RNA below the limit of quantification (BLoQ) by the Abbott RealTime HIV-1 Assay (<40 copies/mL) in both treatment groups.
Time Frame: Immediate Switch to MK-1439A arm: Week 24; Delayed Switch to MK-1439A arm: Week 24
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 447 | 223
Percentage of Participants | 92.8 | 93.3
Statistical Analysis 1: Comparison: Immediate Switch Group (ISG) vs Delayed Switch Group (DSG); Test type: Other; Treatment Difference = -0.427, 95% CI 2-sided [-4.591 to 3.738] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA >=50 Copies/mL
Description: The percentage of participants in each arm achieving HIV-1 RNA levels >=50 copies/mL was determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach.
Time Frame: Immediate Switch to MK-1439A arm: Week 48; Delayed Switch to MK-1439A arm: Week 24
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 447 | 223
Percentage of Participants | 1.6 | 1.8
Statistical Analysis 1: Comparison: Immediate Switch Group (ISG) vs Delayed Switch Group (DSG); Test type: Non-Inferiority — DOR/3TC/TDF QD ISG is concluded to be non-inferior to baseline regimen DSG if the lower bound of the 95% CI for the difference in percent response is above -4 percentage points; Treatment Difference = -0.232, 95% CI 2-sided [-2.529 to 2.064] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percentage of Participants Experiencing ≥1 Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to week 24
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 447 | 223
Percentage of Participants | 68.9 | 52.5

11. Secondary Outcome: Percentage of Participants Experiencing ≥1 Serious Adverse Event (SAE)
Description: A serious adverse event is an AE that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs a hospitalization, is a congenital anomaly or birth defect, is a cancer, is associated with an overdose, or is another important medical event. The percentage of participants with any SAE was assessed.
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 447 | 223
Percentage of Participants | 2.9 | 3.6

12. Secondary Outcome: Percentage of Participants Discontinuing From Study Medication Due to an AE(s)
Description: as for outcome 10
Time Frame: Up to Week 24
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Switch Group (ISG) | Delayed Switch Group (DSG)
Number analyzed (Participants) | 447 | 223
Percentage of Participants | 2.5 | 0.4

ADVERSE EVENTS:
Time Frame: Up to ~338 weeks
Description: All cause-mortality was reported on all allocated participants. Serious and non-serious AEs were reported for all allocated participants who received ≥1 dose of study treatment.
Groups:
- ISG Base Study Weeks 0-24; ISG Base Study Weeks 24-48; ISG Study Extension 1; ISG Study Extension 2; ISG Study Extension 3: Participants received continuous antiretroviral therapy with a ritonavir- or cobicistat-boosted protease inhibitor (atazanavir, darunavir, or lopinavir) or cobicistat-boosted elvitegravir or a non nucleoside reverse transcriptase inhibitor (NNRTI) (specifically, efavirenz, nevirapine, or rilpivirine) in combination with 2 (nuceloside/nucleotide reverse transcriptase inhibitors) NRTIs for >=6 months with undetectable HIV-1 RNA switched on Day 1 to MK-1439A single tablet by mouth once daily for 48 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions.
- DSG Base Study Weeks 0-24; DSG Base Study Weeks 24-48; DSG Study Extension 1; DSG Study Extension 2; DSG Study Extension 3: Participants received continuous antiretroviral therapy with a ritonavir- or cobicistat-boosted protease inhibitor (atazanavir, darunavir, or lopinavir) or cobicistat-boosted elvitegravir or a NNRTI (specifically, efavirenz, nevirapine, or rilpivirine) in combination with 2 NRTIs for >=6 months with undetectable HIV-1 RNA will continue on this therapy until Week 24, at which time they switched to MK-1439A single tablet by mouth once daily for 24 weeks in the Base Study and, optionally, for up to an additional 6 years in the Study Extensions.
Arm/Group | ISG Base Study Weeks 0-24 | DSG Base Study Weeks 0-24 | ISG Base Study Weeks 24-48 | DSG Base Study Weeks 24-48 | ISG Study Extension 1 | DSG Study Extension 1 | ISG Study Extension 2 | DSG Study Extension 2 | ISG Study Extension 3 | DSG Study Extension 3
All-Cause Mortality (participants affected / at risk) | 1/450 | 0/223 | 0/427 | 0/209 | 1/398 | 0/202 | 3/303 | 0/154 | 0/84 | 0/43
Serious Adverse Events (participants affected / at risk) | 13/447 | 8/223 | 11/427 | 4/209 | 37/398 | 13/202 | 13/303 | 7/154 | 3/84 | 1/43
Other Adverse Events (participants affected / at risk) | 100/447 | 28/223 | 63/427 | 33/209 | 107/398 | 57/202 | 24/303 | 11/154 | 9/84 | 3/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISG Base Study Weeks 0-24 (N=447) | DSG Base Study Weeks 0-24 (N=223) | ISG Base Study Weeks 24-48 (N=427) | DSG Base Study Weeks 24-48 (N=209) | ISG Study Extension 1 (N=398) | DSG Study Extension 1 (N=202) | ISG Study Extension 2 (N=303) | DSG Study Extension 2 (N=154) | ISG Study Extension 3 (N=84) | DSG Study Extension 3 (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shigella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISG Base Study Weeks 0-24 (N=447) | DSG Base Study Weeks 0-24 (N=223) | ISG Base Study Weeks 24-48 (N=427) | DSG Base Study Weeks 24-48 (N=209) | ISG Study Extension 1 (N=398) | DSG Study Extension 1 (N=202) | ISG Study Extension 2 (N=303) | DSG Study Extension 2 (N=154) | ISG Study Extension 3 (N=84) | DSG Study Extension 3 (N=43)
Diarrhoea (Gastrointestinal disorders) | 20 (21) | 5 (5) | 13 (13) | 9 (10) | 18 (20) | 11 (14) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 6 (6) | 7 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 33 (34) | 12 (14) | 19 (21) | 9 (10) | 51 (68) | 29 (54) | 5 (5) | 2 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 5 (5) | 8 (9) | 3 (5) | 21 (23) | 4 (4) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4) | 16 (16) | 1 (1) | 21 (22) | 9 (11) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 29 (32) | 5 (5) | 11 (11) | 14 (14) | 22 (24) | 13 (16) | 2 (3) | 3 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT02397096/Prot_SAP_001.pdf